CLINICAL TRIAL: NCT04465526
Title: The Influence of Coronary Chronic Total Occlusion on Myocardial Perfusion on Dual-energy Computed Tomography (COPACABANA Trial)
Brief Title: The Influence of Coronary Chronic Total Occlusion on Myocardial Perfusion on Computed Tomography
Acronym: COPACABANA
Status: Completed | Type: Observational
Sponsor: National Institute of Cardiology, Warsaw, Poland (Other)
Responsible Party: Sponsor
Other Study IDs: 2.31/III/2020
Record Dates: First submitted 2020-07-09; First posted 2020-07-10 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2023-12

CONDITIONS: Coronary Occlusion; Myocardial Ischemia; Myocardial Perfusion Imaging; Percutaneous Coronary Intervention
MeSH Terms: conditions — Coronary Occlusion; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: computed tomography perfusion imaging — The new-generation dual-source computed tomography scanner Somatom® Force will be used for all CTP studies. Myocardial perfusion will be evaluated in a stress dynamic CT protocol. The scan range will be determined based on a low-dose non-contrast scan. Subsequently, regadenoson will be administered intravenously at a single dose of 0.4 mg, and followed after 50 seconds delay by 35 mL of the iodinated contrast agent (iohexol, concentration 350 mg I/mL) injected at the flow rate of 5 mL/s. Finally, low-dose non-contrast dual-energy CT scan will be performed 5-6 min after the dynamic scan to assess late enhancement of the myocardium.

SUMMARY:
The COPACABANA study is designed as a single-centre, open, prospective trial aimed to assess the influence of coronary chronic total occlusion (CTO) on downstream myocardial ischemia via the novel computed tomography perfusion (CTP) imaging technique. To this end, consecutive patients with CTO of a major coronary artery scheduled to undergo percutaneous recanalization of occluded coronary artery based on clinical grounds, will undergo stress CTP using state-of-the-art dual-energy CT scanner at 2 time points (before and 3 months after successful restoration of flow in the CTO vessel).

ELIGIBILITY:
Inclusion Criteria:

* delivery of an informed consent and compliance with study protocol
* persistent angina pectoris (CCS class ≥2) refractory to optimal medical therapy
* CTO of a major coronary artery (left anterior descending artery, right coronary artery, left circumflex artery) of at least 2.5 mm vessel diameter confirmed by invasive angiography
* preserved left ventricular ejection fraction (>50%) on echocardiography or cardiac magnetic resonance with preserved contractility in the CTO territory (normokinesia and/or hypokinesia)

Exclusion Criteria:

* unstable angina and/or myocardial infarction
* prior myocardial infarction within 4 weeks before study enrolment
* occurrence of myocardial infarction and/or unplanned revascularization between the index procedure and post-procedural CTP study
* impaired renal function (eGFR ≤45 ml/min/m2)
* contraindications to antiplatelet therapy and/or heparin
* other contraindications to CTP (pregnancy, allergy to contrast media or pharmacologic stress agents, tachyarrhythmia, claustrophobia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We intend to include 30 consecutive patients with chronic total occlusion of a major coronary artery and preserved left ventricular ejection fraction (>50%) referred for percutaneous recanalization attempt based on clinical grounds.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of stress computed tomography perfusion imaging for myocardial ischemia assessment in patients with a coronary chronic total occlusion | 1 day
  Feasibility of a fast, reliable and safe evaluation of myocardial ischemia in patients with CTO using state-of-the-art computed tomography scanner (SOMATOM® Force) with a dual-energy stress myocardial perfusion imaging protocol in order to obtain in-depth knowledge of the underlying conditions and characteristics of this phenomenon.
Evaluation of myocardial ischemia using stress computed tomography perfusion imaging in patients with a coronary chronic total occlusion | 1 day
  Qualitative and quantitative assessment of myocardial ischemia using stress computed tomography perfusion imaging in patients with a coronary chronic total occlusion.

SECONDARY OUTCOMES:
Change in myocardial perfusion between baseline (pre-procedural) and follow-up (post-procedural) stress computed tomography perfusion study after successful recanalization of the chronically occluded coronary artery | 1 day and 3 months
  Qualitative and quantitative assessment of the change in myocardial perfusion between baseline (pre-procedural) and follow-up (post-procedural) stress computed tomography perfusion study after successful recanalization of the chronically occluded coronary artery.
Radiation dose associated with computed tomography perfusion study in patients with a coronary chronic total occlusion | 1 day and 3 months
  Radiation dose associated with computed tomography perfusion study in patients with a coronary chronic total occlusion undergoing percutaneous recanalization attempt.
Contrast volume associated with computed tomography perfusion study in patients with a coronary chronic total occlusion | 1 day and 3 months
  Contrast volume associated with computed tomography perfusion study in patients with a coronary chronic total occlusion undergoing percutaneous recanalization attempt.

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Cardiology, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kwiecinski J, Oleksiak A, Kruk M, Zysk A, Debski A, Knaapen P, Schumacher SP, Barbero U, Witkowski A, Kepka C, Opolski MP. Computed tomography perfusion and angiography in patients with chronic total occlusion undergoing percutaneous coronary intervention. Atherosclerosis. 2023 Sep;381:117174. doi: 10.1016/j.atherosclerosis.2023.06.080. Epub 2023 Jun 25. PMID 37400307